CLINICAL TRIAL: NCT05428917
Title: Evaluation of the Impact of Laterality on Cerebral Activation During a Motor Task of the Upper Limb Using fNIRS Technology in Healthy Subjects
Brief Title: Evaluation of the Impact of Laterality on Cerebral Activation During a Motor Task of the Upper Limb in Healthy Subjects
Acronym: Lateralinirs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRO-2021-13
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: Laterality; motor task; cerebral activation; near infrared spectroscopy

STUDY DESIGN:
Intervention Model Description: 60 healthy subjects (30 left handed and 30 right handed) will be recruited and will carry out the acquisition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Near infrared spectroscopy (Experimental): This method allows (like fMRI) to study cerebral neurovascular coupling. It is based on the fact that an activated brain region increases its local blood flow. Oxygenated (HbO) and deoxygenated (HbR) hemoglobin absorb infrared light and it is then possible to identify the cerebral cortical regions involved in a given task. This technique therefore makes it possible to study cerebral activation under more ecological conditions than fMRI and is thus particularly suitable for exploring rehabilitation techniques.
  Interventions: Behavioral: Simple task; Behavioral: complex task

INTERVENTIONS:
Behavioral: Simple task — The subject is seated on a chair facing a table, both hands resting on the table.
  The subject is asked, for each block of 20 seconds, to perform flexion / extension movements of the fingers of the left hand at 0.5 Hz.
Behavioral: complex task — The subject is seated on a chair facing a table, both hands resting on the table.
  The subject is asked, for each block of 20 seconds, to perform an exercise based on the nine hole peg test

SUMMARY:
The aim of this study is to investigate the differences in brain activation in healthy subjects during motor tasks, depending on the laterality of the subject, the laterality of the task and the complexity of the task. It seems that the laterality of activation is less marked in left-handed people, when using the non-dominant hand and when performing a complex task. The objective of this study is to highlight profiles of subject and modality of use of the hand with a specific lateralization of cerebral activation.

DETAILED DESCRIPTION:
Stroke frequently leads to upper limb deficit. The recovery of motor skills depends on many factors including laterality. The literature shows that cerebral activation during motor tasks differs depending on whether one is right-handed or left-handed and whether one uses the dominant hand or not. These differences probably lead to different recovery mechanisms depending on the side of the lesion and the laterality. An imaging technique is particularly suitable for exploring these different mechanisms: fNIRS (Functional Near Infra Red Spectroscopy). This method allows (like fMRI) to study cerebral neurovascular coupling. It is based on the fact that an activated brain region increases its local blood flow. Oxygenated (HbO) and deoxygenated (HbR) hemoglobin absorb infrared light and it is then possible to identify the cerebral cortical regions involved in a given task. This technique therefore makes it possible to study cerebral activation under more ecological conditions than fMRI and is thus particularly suitable for exploring rehabilitation techniques.

This research aims to study and compare in healthy subjects, using an fNIRS apparatus, the brain regions involved in the performance of different motor tasks according to the laterality of the task and the subject.

The investigations will be carried out by the principal investigator or by specialized technicians from the neurology functional exploration department.

Stroke frequently leads to upper limb deficit. The recovery of motor skills depends on many factors including laterality. The literature shows that cerebral activation during motor tasks differs depending on whether one is right-handed or left-handed and whether one uses the dominant hand or not. These differences probably lead to different recovery mechanisms depending on the side of the lesion and the laterality. An imaging technique is particularly suitable for exploring these different mechanisms: fNIRS (Functional Near Infra Red Spectroscopy). This method allows (like fMRI) to study cerebral neurovascular coupling. It is based on the fact that an activated brain region increases its local blood flow. Oxygenated (HbO) and deoxygenated (HbR) hemoglobin absorb infrared light and it is then possible to identify the cerebral cortical regions involved in a given task. This technique therefore makes it possible to study cerebral activation under more ecological conditions than fMRI and is thus particularly suitable for exploring rehabilitation techniques.

This research aims to study and compare in healthy subjects, using an fNIRS apparatus, the brain regions involved in the performance of different motor tasks according to the laterality of the task and the subject.

The investigations will be carried out by the principal investigator or by specialized technicians from the neurology functional exploration department.

The acquisition has a duration of 25 minutes, it begins with a rest period of 120 seconds, which corresponds to the baseline. Four different tasks are performed during the acquisition for each subject:

* Simple task right hand (SD)
* Simple task left hand (SG)
* Complex task right hand (CD)
* Complex stain left hand (CG)

The design is a block design, each task, which has a duration of 20 seconds, is carried out 8 times per acquisition. There is therefore a total of 32 tasks whose order will be randomized.

For simple tasks, movements are performed at a frequency of 0.5 Hz which appears to be the optimal frequency for observing cortical activation using a metronome.

Between periods of movement, the subject is in a rest position for a period from 15 to 25 seconds.

Instructions are given verbally at the start of each phase. After recruiting the subjects, the study investigator will check the inclusion and exclusion criteria.

If the subject can integrate the protocol, the acquisition will then be planned.

On the day of the acquisition, the fNIRS acquisition helmet (Brite MKII) will be installed by a specialist technician and instructions will be given. The recording is then made.

ELIGIBILITY:
Inclusion Criteria:

* Subject from 18 to 60 years old
* Sufficient command of the French language to understand the instructions
* No known neurological medical history
* Benefiting from social security coverage
* For right-handed subjects: Edinburgh laterality test QL> 40
* For left-handed subjects: Edinburgh laterality test QL< -40

Exclusion Criteria:

* Known allergy to components of the fNIRS device : neoprene

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Laterality index using t values | Minutes 25
  Compare the asymmetry of activation of the sensorimotor cortex during a complex motor task on the dominant side between right-handers and left-handers.

SECONDARY OUTCOMES:
concentration of oxyhemoglobin measured with fnirs device | Minutes 25
  Assess the effect of task complexity and the effect of using the dominant or non-dominant side
concentration of deoxyhemoglobin measured with fnirs device | minutes 25
  Assess the effect of task complexity and the effect of using the dominant or non-dominant side

CONTACTS AND LOCATIONS:
Overall Officials: Julien BONNAL, Principal Investigator — Regional Hospital Center of ORLEANS
Locations (1):
- Regional Hospital Center of ORLEANS, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartur G, Pratt H, Dickstein R, Frenkel-Toledo S, Geva A, Soroker N. Electrophysiological manifestations of mirror visual feedback during manual movement. Brain Res. 2015 May 5;1606:113-24. doi: 10.1016/j.brainres.2015.02.029. Epub 2015 Feb 23. PMID 25721791
- [Background] Bondi D, Prete G, Malatesta G, Robazza C. Laterality in Children: Evidence for Task-Dependent Lateralization of Motor Functions. Int J Environ Res Public Health. 2020 Sep 15;17(18):6705. doi: 10.3390/ijerph17186705. PMID 32942557
- [Background] Harris JE, Eng JJ. Individuals with the dominant hand affected following stroke demonstrate less impairment than those with the nondominant hand affected. Neurorehabil Neural Repair. 2006 Sep;20(3):380-9. doi: 10.1177/1545968305284528. PMID 16885424
- [Background] Ludemann-Podubecka J, Bosl K, Theilig S, Wiederer R, Nowak DA. The Effectiveness of 1 Hz rTMS Over the Primary Motor Area of the Unaffected Hemisphere to Improve Hand Function After Stroke Depends on Hemispheric Dominance. Brain Stimul. 2015 Jul-Aug;8(4):823-30. doi: 10.1016/j.brs.2015.02.004. Epub 2015 Mar 16. PMID 25828427
- [Background] Duboc V, Dufourcq P, Blader P, Roussigne M. Asymmetry of the Brain: Development and Implications. Annu Rev Genet. 2015;49:647-72. doi: 10.1146/annurev-genet-112414-055322. Epub 2015 Oct 6. PMID 26442849
- [Background] Grabowska A, Gut M, Binder M, Forsberg L, Rymarczyk K, Urbanik A. Switching handedness: fMRI study of hand motor control in right-handers, left-handers and converted left-handers. Acta Neurobiol Exp (Wars). 2012;72(4):439-51. doi: 10.55782/ane-2012-1914. PMID 23377273
- [Background] Jin SH, Lee SH, Yang ST, An J. Hemispheric asymmetry in hand preference of right-handers for passive vibrotactile perception: an fNIRS study. Sci Rep. 2020 Aug 7;10(1):13423. doi: 10.1038/s41598-020-70496-y. PMID 32770115
- [Background] Kim SG, Ashe J, Hendrich K, Ellermann JM, Merkle H, Ugurbil K, Georgopoulos AP. Functional magnetic resonance imaging of motor cortex: hemispheric asymmetry and handedness. Science. 1993 Jul 30;261(5121):615-7. doi: 10.1126/science.8342027.
- [Background] Lee SH, Jin SH, An J. The difference in cortical activation pattern for complex motor skills: A functional near- infrared spectroscopy study. Sci Rep. 2019 Oct 1;9(1):14066. doi: 10.1038/s41598-019-50644-9. PMID 31575954
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] O'Regan L, Serrien DJ. Individual Differences and Hemispheric Asymmetries for Language and Spatial Attention. Front Hum Neurosci. 2018 Oct 4;12:380. doi: 10.3389/fnhum.2018.00380. eCollection 2018. PMID 30337864
- [Background] Solodkin A, Hlustik P, Noll DC, Small SL. Lateralization of motor circuits and handedness during finger movements. Eur J Neurol. 2001 Sep;8(5):425-34. doi: 10.1046/j.1468-1331.2001.00242.x. PMID 11554905
- [Background] Vingerhoets G, Acke F, Alderweireldt AS, Nys J, Vandemaele P, Achten E. Cerebral lateralization of praxis in right- and left-handedness: same pattern, different strength. Hum Brain Mapp. 2012 Apr;33(4):763-77. doi: 10.1002/hbm.21247. Epub 2011 Apr 15. PMID 21500314